CLINICAL TRIAL: NCT05932277
Title: A Phase 1 Open-label Study to Assess the Effect of BMS-986419 on the Single Dose Pharmacokinetics of Probe Substrates (Caffeine, Bupropion, Flurbiprofen, Omeprazole, Midazolam, and Fexofenadine) in Healthy Participants
Brief Title: A Study to Assess the Effect of BMS-986419 on the Single Dose Drug Levels of Probe Substrates in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN007-1000
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: healthy; pharmacokinetics; BMS-986419
MeSH Terms: interventions — Caffeine; Bupropion; Flurbiprofen; Omeprazole; Midazolam; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cocktail Probe Substrates + BMS-986419 (Experimental)
  Interventions: Drug: BMS-986419; Drug: Caffeine; Drug: Bupropion; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam; Drug: Fexofenadine

INTERVENTIONS:
Drug: BMS-986419 — Specified dose on specified days
Drug: Caffeine — Specified dose on specified days
Drug: Bupropion — Specified dose on specified days
Drug: Flurbiprofen — Specified dose on specified days
Drug: Omeprazole — Specified dose on specified days
Drug: Midazolam — Specified dose on specified days
Drug: Fexofenadine — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the effect of BMS-986419 on the pharmacokinetics (PK) of single doses of caffeine (CYP1A2 substrate), bupropion (CYP2B6 substrate), midazolam (CYP3A4 substrate), flurbiprofen (CYP2C9 substrate), omeprazole (CYP2C19 substrate), and fexofenadine (P-gp substrate), in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants without clinically significant deviation from normal in medical history, physical examination (PE), electrocardiogram (ECG), and clinical laboratory determinations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in (Day -1).
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive, and total body weight ≥ 50 kg. BMI may be rounded.

Exclusion Criteria:

* Any significant acute or chronic medical conditions or any significant acute or chronic medical illness as determined by the investigator
* Any major surgery within 30 days of study intervention administration, such as gastrointestinal surgery that could impact the absorption of study intervention

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 25
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to Day 25
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 25

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 25
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to Day 25
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 25
Number of participants with Adverse Events (AEs) | Up to 28 days after last dose
Number of participants with Serious Adverse Events (SAEs) | Up to 28 days after last dose
Number of participants with AEs leading to discontinuation | Up to 28 days after last dose
Number of participants with vital sign abnormalities | Up to Day 25
Number of participants with 12-lead ECG assessment abnormalities | Up to Day 25
Number of participants with physical examination abnormalities | Up to Day 25
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 25
Number of participants with clinical laboratory abnormalities | Up to Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome